CLINICAL TRIAL: NCT01796652
Title: A Randomized Controlled Trial of Home Monitoring Versus Hospitalization in Mild Non-Alcoholic Acute Interstitial Pancreatitis
Brief Title: Home Treatment of Acute Pancreatitis
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Ali Tüzün İnce, Asc Prof, Bezmialem Vakif University
Other Study IDs: B.30.2.BAV.0.05.05/374
Record Dates: First submitted 2013-02-19; First posted 2013-02-22 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Acute Pancreatitis
Keywords: Acute interstitial pancreatitis; Home therapy
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Home and hospital treatment groups: Patients were randomized into either home or hospital groups after a brief hospitalization(≤24 hours. Hospital patients were followed 5 days in hospital.Home patients were visited on 2nd,3rd and 5th days by a staff nurse and the vital signs, symptoms, and general condition were recorded and transmitted back to the attending physician. On the 7th, 14th and 30th days, the home and hospital group patients were requested to return for a follow-up clinic visit at Bezmialem, at which time an assessment of their symptoms, physical examination, and laboratory evaluation was conducted.

SUMMARY:
Acute pancreatitis (AP) is considered a disease requiring in-hospital treatment. We studied the feasibility of home management in AP.The aim of study was to compare 30 day readmission rates in patients with mild non-alcoholic acute pancreatitis (NAAP) randomized to home monitoring versus hospitalization.

DETAILED DESCRIPTION:
Between 11/11-5/12, 84 patients with mild NAAP were randomized to home or hospital groups after a short (≤24 hours) hospital stay. AP was defined as ≥2 or more of the following: characteristic abdominal pain, amylase and/or lipase ≥3X the upper limit of normal, and/or imaging findings. Patients with an Imrie's score ≤5 and a harmless acute pancreatitis score (HAPS) ≤2 were included. Patients in both groups received intravenous lactated Ringer for 3 days and pain was treated with intramuscular diclofenac. A nurse visited all patients in the home group on the 2nd, 3rd and 5th day. All patients recalled for follow-up on the 7th, 14th, and 30th days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AP based on 2 out of 3 findings: characteristic abdominal pain, amylase and/or lipase levels ≥3 times the upper limit of normal, and/or abdominal imaging demonstrating changes of acute pancreatitis
* Presentation within 48 hours of symptom onset
* Imrie's scores of ≤5 and HAP score ≤2 within 24 hours of presentation to the hospital
* Lack of hemoconcentration (hematocrit ≥44%) on presentation since hemoconcentration has been shown to be a risk factor for pancreatic necrosis.

Exclusion Criteria:

* The presence of organ failure by the Atlanta criteria on the first day of presentation
* The presence of clinical signs and/or symptoms of sepsis
* Alcoholic acute pancreatitis
* A history of abdominal imaging demonstrating a dilated pancreatic duct and/or pancreatic calcifications
* Coagulopathy (international normalized ratio >1, and/or platelet count <50,000/mm3
* Comorbidities requiring hospitalization regardless of the presence of AP e.g. acute myocardial infarction, malignancy, cirrhosis, chronic kidney disease, and chronic pulmonary disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mild acute non-alhololic patients managed in home.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study was the 30 day hospital readmission rate. | 30 days
  30 day hospital readmission of home and hospital groups of patients were evaluated.

SECONDARY OUTCOMES:
Other outcomes evaluated included the duration of abdominal pain and time to resumption of an oral diet, both measured in hours from the time of presentation. | hours
  Elaboration time of abdominal pain in home and hospital group patients as hour from the admission time to ICU.
  Time to resumption of an oral diet measured from the time of presentation.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Şentürk, Prof., Principal Investigator — Bezmialem Vakıf University Hospital, Gastroenterology Clinic
Locations (1):
- Bezmialem Vakıf University Hospital, Gastroenterology Clinic, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Whitlock TL, Repas K, Tignor A, Conwell D, Singh V, Banks PA, Wu BU. Early readmission in acute pancreatitis: incidence and risk factors. Am J Gastroenterol. 2010 Nov;105(11):2492-7. doi: 10.1038/ajg.2010.234. Epub 2010 Jun 8. PMID 20531398
- [Background] Rodriguez-Cerrillo M, Poza-Montoro A, Fernandez-Diaz E, Inurrieta-Romero A, Matesanz-David M. Home treatment of patients with acute cholecystitis. Eur J Intern Med. 2012 Jan;23(1):e10-3. doi: 10.1016/j.ejim.2011.07.012. Epub 2011 Aug 27. PMID 22153541
- [Background] van Baal MC, Besselink MG, Bakker OJ, van Santvoort HC, Schaapherder AF, Nieuwenhuijs VB, Gooszen HG, van Ramshorst B, Boerma D; Dutch Pancreatitis Study Group. Timing of cholecystectomy after mild biliary pancreatitis: a systematic review. Ann Surg. 2012 May;255(5):860-6. doi: 10.1097/SLA.0b013e3182507646. PMID 22470079
- [Background] Andersson B, Pendse ML, Andersson R. Pancreatic function, quality of life and costs at long-term follow-up after acute pancreatitis. World J Gastroenterol. 2010 Oct 21;16(39):4944-51. doi: 10.3748/wjg.v16.i39.4944. PMID 20954281
- [Derived] Ince AT, Senturk H, Singh VK, Yildiz K, Danalioglu A, Cinar A, Uysal O, Kocaman O, Baysal B, Gurakar A. A randomized controlled trial of home monitoring versus hospitalization for mild non-alcoholic acute interstitial pancreatitis: a pilot study. Pancreatology. 2014 May-Jun;14(3):174-8. doi: 10.1016/j.pan.2014.02.007. Epub 2014 Mar 14. PMID 24854612